CLINICAL TRIAL: NCT01403948
Title: A Phase I, Open-Label, Dose-Escalation Trial With BI 836826 in Patients With Relapsed or Refractory Non-Hodgkin Lymphoma of B Cell Origin
Brief Title: BI 836826 Dose Escalation in Patients With Relapsed or Refractory Non-Hodgkin Lymphoma (NHL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1270.2; 2010-024456-29 (EudraCT Number)
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — BI 836826

ARMS (1):
- Patients with relapsed or refractory NHL (Experimental): Adult patients with relapsed or refractory non-Hodgkin lymphoma of B cell origin after at least two prior treatments
  Interventions: Drug: BI 836826

INTERVENTIONS:
Drug: BI 836826 — Monotherapy with BI 836826 at escalating dose levels administered as an intravenous infusion

SUMMARY:
The purpose is to investigate the maximum tolerated dose (MTD), safety and tolerability, pharmacokinetics and efficacy of BI 836826 monotherapy in patients with relapsed or refractory non-Hodgkin lymphoma with at least prior treatments.

ELIGIBILITY:
Inclusion criteria:

1. Patients with relapsed or refractory non-Hodgkin lymphoma of B cell origin (mature B cell lymphoma according to WHO) not considered candidates for intensive anti-lymphoma therapy
2. Patients must have either aggressive NHL and received at least one prior anti-CD20 containing immunochemotherapy or indolent NHL and received anti-CD20 therapy and at least two prior therapies
3. Measurable disease on computed tomography (CT) scan with involvement of one clearly demarcated lesion =2 cm or two or more clearly demarcated lesions of >1.5 cm at longest diameter (this criterion applies only for the expansion cohort)
4. Relapse or progression of disease with an indication for therapy as per investigator's judgement
5. Life expectancy of =3 months
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1

Exclusion criteria:

1. Primary central nervous system (CNS) lymphoma or known CNS involvement
2. Prior history of malignancy other than a mature B cell neoplasm according to WHO classification (except basal cell or squamous cell carcinoma of the skin, or carcinoma in situ of the uterine cervix or breast treated with curative therapy) unless the subject has been free of disease and without treatment for at least 5 years
3. Last chemotherapy <4 weeks prior to visit 1
4. Last anti-CD20 therapy (non-radiolabelled) <4 weeks prior to visit 1
5. Last corticosteroid <2 weeks prior to visit 1 unless the dose is less or equal of 10 mg/day prednisolone or equivalent
6. High-dose therapy with stem cell support <6 months prior to visit 1
7. Radio-immunotherapy <3 months prior to visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (12):
- France (2):
  - INS Paoli-Calmettes, Marseille
  - HOP Lyon Sud, Pierre-Bénite
- Germany (8):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsmedizin Göttingen, Georg-August-Universität, Göttingen
  - Asklepios Klinik St. Georg, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Ulm, Ulm
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Kroschinsky F, Middeke JM, Janz M, Lenz G, Witzens-Harig M, Bouabdallah R, La Rosee P, Viardot A, Salles G, Kim SJ, Kim TM, Ottmann O, Chromik J, Quinson AM, von Wangenheim U, Burkard U, Berk A, Schmitz N. Phase I dose escalation study of BI 836826 (CD37 antibody) in patients with relapsed or refractory B-cell non-Hodgkin lymphoma. Invest New Drugs. 2020 Oct;38(5):1472-1482. doi: 10.1007/s10637-020-00916-3. Epub 2020 Mar 14. PMID 32172489

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label trial with a dose-escalation phase according to a modified 3+3 design.
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be entered to trial drug if any of the specific entry criteria was violated.
Groups:
- BI 836826 1 mg iv (Caucasian Patients): BI 836826 1 milligram (mg) was administered as an intravenous (iv) infusion anytime in day (preferably morning hours) in caucasian patients with relapsed or refractory non-hodgkin lymphoma of B cell origin.
  Each course was to comprise 4 administrations at weekly intervals, followed by 27 days of observation after last administration. The duration of the 2 first courses was 7 weeks each and the duration of the 3rd course was 12 weeks. The maximum duration of the treatment and observation/rest periods was 26 weeks.
- BI 836826 3 mg iv (Caucasian Patients): BI 836826 3 mg was administered as an intravenous infusion anytime in day (preferably morning hours) in caucasian patients with relapsed or refractory non-hodgkin lymphoma of B cell origin.
  Each course was to comprise 4 administrations at weekly intervals, followed by 27 days of observation after last administration. The duration of the 2 first courses was 7 weeks each and the duration of the 3rd course was 12 weeks. The maximum duration of the treatment and observation/rest periods was 26 weeks.
- BI 836826 9 mg iv (Caucasian Patients): BI 836826 9 mg was administered as an intravenous infusion anytime in day (preferably morning hours) in caucasian patients with relapsed or refractory non-hodgkin lymphoma of B cell origin.
  Each course was to comprise 4 administrations at weekly intervals, followed by 27 days of observation after last administration. The duration of the 2 first courses was 7 weeks each and the duration of the 3rd course was 12 weeks. The maximum duration of the treatment and observation/rest periods was 26 weeks.
- BI 836826 25 mg iv (Caucasian Patients): BI 836826 25 mg was administered as an intravenous infusion anytime in day (preferably morning hours) in caucasian patients with relapsed or refractory non-hodgkin lymphoma of B cell origin.
  Each course was to comprise 4 administrations at weekly intervals, followed by 27 days of observation after last administration. The duration of the 2 first courses was 7 weeks each and the duration of the 3rd course was 12 weeks. The maximum duration of the treatment and observation/rest periods was 26 weeks.
- BI 836826 50 mg iv (Caucasian Patients): BI 836826 50 mg was administered as an intravenous infusion anytime in day (preferably morning hours) in caucasian patients with relapsed or refractory non-hodgkin lymphoma of B cell origin.
  Each course was to comprise 4 administrations at weekly intervals, followed by 27 days of observation after last administration. The duration of the 2 first courses was 7 weeks each and the duration of the 3rd course was 12 weeks. The maximum duration of the treatment and observation/rest periods was 26 weeks.
- BI 836826 50mg iv (Korean Patients): BI 836826 50 mg was administered as an intravenous infusion anytime in day (preferably morning hours) in korean patients with relapsed or refractory non-hodgkin lymphoma of B cell origin.
  Each course was to comprise 4 administrations at weekly intervals, followed by 27 days of observation after last administration. The duration of the 2 first courses was 7 weeks each and the duration of the 3rd course was 12 weeks. The maximum duration of the treatment and observation/rest periods was 26 weeks.
- BI 836826 100 mg iv (Caucasian Patients): BI 836826 100 mg was administered as an intravenous infusion anytime in day (preferably morning hours) in caucasian patients with relapsed or refractory non-hodgkin lymphoma of B cell origin.
  Each course was to comprise 4 administrations at weekly intervals, followed by 27 days of observation after last administration. The duration of the 2 first courses was 7 weeks each and the duration of the 3rd course was 12 weeks. The maximum duration of the treatment and observation/rest periods was 26 weeks.
- BI 836826 100 mg iv (Korean Patients): BI 836826 100 mg was administered as an intravenous infusion anytime in day (preferably morning hours) in korean patients with relapsed or refractory non-hodgkin lymphoma of B cell origin.
  Each course was to comprise 4 administrations at weekly intervals, followed by 27 days of observation after last administration. The duration of the 2 first courses was 7 weeks each and the duration of the 3rd course was 12 weeks. The maximum duration of the treatment and observation/rest periods was 26 weeks.
- BI 836826 150 mg iv (Caucasian Patients): BI 836826 150 mg was administered as an intravenous infusion anytime in day (preferably morning hours) in caucasian patients with relapsed or refractory non-hodgkin lymphoma of B cell origin.
  Each course was to comprise 4 administrations at weekly intervals, followed by 27 days of observation after last administration. The duration of the 2 first courses was 7 weeks each and the duration of the 3rd course was 12 weeks. The maximum duration of the treatment and observation/rest periods was 26 weeks.
- BI 836826 200 mg iv (Caucasian Patients): BI 836826 200 mg was administered as an intravenous infusion anytime in day (preferably morning hours) in caucasian patients with relapsed or refractory non-hodgkin lymphoma of B cell origin.
  Each course was to comprise 4 administrations at weekly intervals, followed by 27 days of observation after last administration. The duration of the 2 first courses was 7 weeks each and the duration of the 3rd course was 12 weeks. The maximum duration of the treatment and observation/rest periods was 26 weeks.
Period: Overall Study
Arm/Group | BI 836826 1 mg iv (Caucasian Patients) | BI 836826 3 mg iv (Caucasian Patients) | BI 836826 9 mg iv (Caucasian Patients) | BI 836826 25 mg iv (Caucasian Patients) | BI 836826 50 mg iv (Caucasian Patients) | BI 836826 50mg iv (Korean Patients) | BI 836826 100 mg iv (Caucasian Patients) | BI 836826 100 mg iv (Korean Patients) | BI 836826 150 mg iv (Caucasian Patients) | BI 836826 200 mg iv (Caucasian Patients)
Started | 1 | 4 | 3 | 4 | 6 | 7 | 6 | 4 | 6 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 4 | 3 | 4 | 6 | 7 | 6 | 4 | 6 | 7
Not completed — Progressive disease | 0 | 2 | 2 | 4 | 2 | 6 | 2 | 4 | 5 | 5
Not completed — Other Adverse Event (Other than DLT) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Refused cont. medication | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — other than above | 1 | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): Treated set (TS) consists of all patients who received at least 1 dose of BI 836826.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 836826 1 mg iv (Caucasian Patients) | BI 836826 3 mg iv (Caucasian Patients) | BI 836826 9 mg iv (Caucasian Patients) | BI 836826 25 mg iv (Caucasian Patients) | BI 836826 50 mg iv (Caucasian Patients) | BI 836826 50mg iv (Korean Patients) | BI 836826 100 mg iv (Caucasian Patients) | BI 836826 100 mg iv (Korean Patients) | BI 836826 150 mg iv (Caucasian Patients) | BI 836826 200 mg iv (Caucasian Patients) | Total
Number analyzed (Participants) | 1 | 4 | 3 | 4 | 6 | 7 | 6 | 4 | 6 | 7 | 48
Age, Continuous [Median (Full Range); unit: Years] | 75.0 [75 to 75] | 75.0 [71 to 83] | 61.0 [57 to 69] | 69.5 [46 to 78] | 74.5 [45 to 76] | 57.0 [27 to 79] | 69.0 [56 to 80] | 70.0 [58 to 79] | 66.0 [55 to 73] | 68.0 [25 to 83] | 68.5 [25 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 1 | 2 | 4 | 2 | 3 | 1 | 3 | 18
  Male | 1 | 4 | 1 | 3 | 4 | 3 | 4 | 1 | 5 | 4 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethinicity was not captured in this trial.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 4 | 0 | 0 | 11
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    White | 1 | 4 | 3 | 4 | 6 | 0 | 6 | 0 | 4 | 5 | 33
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Maximum Tolerated Dose (MTD) Based on the Occurrence of Dose-limiting Toxicity (DLT) in First Cycle in Caucasian Patients
Description: The primary objective of the dose-escalation part of this study was to determine the MTD of BI 836826 in caucasian patients. The MTD was to be defined on the basis of DLTs observed during the first 2 weeks of the 1st treatment course. In case of a delay of the second administration, evaluation of DLT was to be prolonged to 7 days after the second administration.. A DLT was defined as any drug-related non-haematological Adverse event (AE) of Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 or higher, except Infusion-related reaction (IRRs) associated with the administration of BI 836826.
Time Frame: From the first administration of trial medication to 7 days after the second administration, upto 36 days
Population: Treated Set
Measure: Number; unit: Milligram (mg)
Groups:
- BI 836826: Caucasian patients were treated in the dose-escalation phase with BI 836826 as an intravenous infusion until the patient met criteria for stopping study medication during the MTD evaluation period. The duration of the 2 first courses was 7 weeks each and the duration of the 3rd course was 12 weeks. The maximum duration of the treatment and observation/rest periods was 26 weeks.
Arm/Group | BI 836826
Number analyzed (Participants) | 37
Milligram (mg) | 100

2. Primary Outcome: Number of Subjects With Dose Limiting Toxicities (DLT) in First Cycle in Caucasian Patients
Description: Number of subjects with Dose Limiting Toxicities (DLT) in first Cycle during the MTD evaluation period in caucasian patients with relapsed or refractory Non-Hodgkin lymphoma (NHL).
Time Frame: From the first administration of trial medication to 7 days after the second administration, up to 36 days
Population: Treated Set
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836826 1 mg iv (Caucasian Patients) | BI 836826 3 mg iv (Caucasian Patients) | BI 836826 9 mg iv (Caucasian Patients) | BI 836826 25 mg iv (Caucasian Patients) | BI 836826 50 mg iv (Caucasian Patients) | BI 836826 100 mg iv (Caucasian Patients) | BI 836826 150 mg iv (Caucasian Patients) | BI 836826 200 mg iv (Caucasian Patients)
Number analyzed (Participants) | 1 | 4 | 3 | 4 | 6 | 6 | 6 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1

3. Secondary Outcome: Tumour Size Reduction
Description: Tumour size reduction (lymph nodes, spleen, & liver nodules) defined as best percentage change from baseline in sum of products of diameter (SPD). Negative value represents decrease in tumour size, & positive value represents an increase in size. The tumour size of lymph nodes was to be measured as SPD of 2 perpendicular dimensions for up to 6 indicator lesions identified at baseline CT scan. Spleen & liver were to be described if considered enlarged at baseline by physical examination or CT scan. If nodules present in spleen &/or liver, was to be measured in 2 perpendicular dimensions. Median, 25th & 75th percentiles are calculated from unadjusted Kaplan-Meier curve for each treatment cohort.
Time Frame: Computed tomography (CT) scan performed at screening, at Week 13, and at Week 25.
Population: Treated set
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | BI 836826 1 mg iv (Caucasian Patients) | BI 836826 3 mg iv (Caucasian Patients) | BI 836826 9 mg iv (Caucasian Patients) | BI 836826 25 mg iv (Caucasian Patients) | BI 836826 50 mg iv (Caucasian Patients) | BI 836826 50mg iv (Korean Patients) | BI 836826 100 mg iv (Caucasian Patients) | BI 836826 100 mg iv (Korean Patients) | BI 836826 150 mg iv (Caucasian Patients) | BI 836826 200 mg iv (Caucasian Patients)
Number analyzed (Participants) | 1 | 4 | 3 | 4 | 6 | 7 | 6 | 4 | 6 | 7
Percentage
  indicator lesions: number analyzed (Participants) | 1 | 3 | 2 | 3 | 4 | 5 | 4 | 3 | 3 | 1
  indicator lesions | -44.74 (NA) — Only one patient has been analysed thus SD is not calculable | 118.42 (183.49) | -0.11 (61.72) | 67.26 (61.78) | -3.72 (10.19) | 28.80 (78.03) | -9.44 (34.49) | 110.88 (41.82) | 60.13 (29.68) | 1.90 (NA) — Only one patient has been analysed thus SD is not calculable
  liver nodules: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  liver nodules |  |  |  |  |  |  |  |  |  | 33.16 (NA) — Only one patient has been analysed thus SD is not calculable
  spleen nodules: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Best Overall Response Based on All Assessment
Description: Best overall response was best response at any of CT scans and investigator assesment (incase the recent CT scan was not available). Response was assessed as follow according to the Standardized or Revised Response Criteria for Malignant Lymphoma from 1999.:
  1. Complete remission (CR)
  2. Complete remission unconfirmed (CRu)
  3. Partial remission (PR)
  4. Stable disease (SD)
  5. progressive disease (PD)
Time Frame: Screening, Week 1, Week 4, Week 7, Week 8, Week 11, Week 14, Week 15, Week 18 and at End of Treatment (EOT)
Population: Treated set
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836826 1 mg iv (Caucasian Patients) | BI 836826 3 mg iv (Caucasian Patients) | BI 836826 9 mg iv (Caucasian Patients) | BI 836826 25 mg iv (Caucasian Patients) | BI 836826 50 mg iv (Caucasian Patients) | BI 836826 50mg iv (Korean Patients) | BI 836826 100 mg iv (Caucasian Patients) | BI 836826 100 mg iv (Korean Patients) | BI 836826 150 mg iv (Caucasian Patients) | BI 836826 200 mg iv (Caucasian Patients)
Number analyzed (Participants) | 1 | 4 | 3 | 4 | 6 | 7 | 6 | 4 | 6 | 7
Participants
  Complete remission | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Complete remission unconfirmed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial remission | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
  Stable disease | 1 | 3 | 2 | 2 | 3 | 3 | 2 | 2 | 0 | 2
  Progressive disease | 0 | 0 | 1 | 2 | 1 | 3 | 0 | 2 | 5 | 4
  Missing | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1

5. Secondary Outcome: Best Overall Response Based on Imaging Data
Description: Best overall response based on imaging data. Response was assessed as follow according to the Standardized or Revised Response Criteria for Malignant Lymphoma from 1999.:
  1. Complete remission
  2. Complete remission unconfirmed
  3. Partial remission
  4. Stable disease:
  5. progressive disease
Time Frame: Computed tomography (CT) scan performed at screening, at Week 13, and at Week 25.
Population: Treated set
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836826 1 mg iv (Caucasian Patients) | BI 836826 3 mg iv (Caucasian Patients) | BI 836826 9 mg iv (Caucasian Patients) | BI 836826 25 mg iv (Caucasian Patients) | BI 836826 50 mg iv (Caucasian Patients) | BI 836826 50mg iv (Korean Patients) | BI 836826 100 mg iv (Caucasian Patients) | BI 836826 100 mg iv (Korean Patients) | BI 836826 150 mg iv (Caucasian Patients) | BI 836826 200 mg iv (Caucasian Patients)
Number analyzed (Participants) | 1 | 4 | 3 | 4 | 6 | 7 | 6 | 4 | 6 | 7
Participants
  Complete remission | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Complete remission unconfirmed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial remission | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Stable disease | 1 | 1 | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 2
  Progressive disease | 0 | 2 | 2 | 4 | 2 | 5 | 2 | 4 | 5 | 4
  Missing | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from first treatment with BI 836826 until disease progression or death from any cause. For disease progression one of the following criteria was required:
  • Any new lesion >1.5 centimeter (cm) in any axis • Increase of ≥50% from nadir in sum of product of diameter of any previously involved nodes or single nodes or the size of hepatic or splenic nodules. A lymph node with a diameter of the short axis of <1 cm had to increase by ≥50% and to a size of 1.5 x 1.5 cm or more than 1.5 cm in the long axis • Increase of ≥50% in the longest diameter of any single previously identified node >1 cm in its short axis. Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve for each treatment cohort.
Time Frame: from first treatment until disease progression or death from any cause, up to 12 months.
Population: Treated set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | BI 836826 1 mg iv (Caucasian Patients) | BI 836826 3 mg iv (Caucasian Patients) | BI 836826 9 mg iv (Caucasian Patients) | BI 836826 25 mg iv (Caucasian Patients) | BI 836826 50 mg iv (Caucasian Patients) | BI 836826 50mg iv (Korean Patients) | BI 836826 100 mg iv (Caucasian Patients) | BI 836826 100 mg iv (Korean Patients) | BI 836826 150 mg iv (Caucasian Patients) | BI 836826 200 mg iv (Caucasian Patients)
Number analyzed (Participants) | 1 | 4 | 3 | 4 | 6 | 7 | 6 | 4 | 6 | 7
days | 352.00 [352.00 to 352.00] | 87.00 [47.00 to NA] — Not calculable due to insufficient number of patients with event | 81.00 [17.00 to NA] — Not calculable due to insufficient number of patients with event | 22.00 [12.00 to 36.00] | 262.00 [85.00 to 262.00] | 27.50 [24.00 to 38.00] | 200.00 [62.00 to 218.00] | 51.50 [39.50 to 88.50] | 34.00 [22.00 to 44.00] | 38.00 [19.00 to NA] — Not calculable due to insufficient number of patients with event

7. Secondary Outcome: Failure Free Survival (FFS)
Description: FFS was defined as the time from first treatment with BI 836826 until objective disease progression, death, or start of next Non-Hodgkin lymphoma (NHL) therapy.For disease progression one of the following criteria was required:
  • Any new lesion >1.5 centimeter (cm) in any axis • Increase of ≥50% from nadir in sum of product of diameter of any previously involved nodes or single nodes or the size of hepatic or splenic nodules. A lymph node with a diameter of the short axis of <1 cm had to increase by ≥50% and to a size of 1.5 x 1.5 cm or more than 1.5 cm in the long axis • Increase of ≥50% in the longest diameter of any single previously identified node >1 cm in its short axis. Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve for each treatment cohort.
Time Frame: from first treatment with BI 836826 until objective disease progression, death, or start of next NHL therapy, up to 12 months.
Population: Treated set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | BI 836826 1 mg iv (Caucasian Patients) | BI 836826 3 mg iv (Caucasian Patients) | BI 836826 9 mg iv (Caucasian Patients) | BI 836826 25 mg iv (Caucasian Patients) | BI 836826 50 mg iv (Caucasian Patients) | BI 836826 50mg iv (Korean Patients) | BI 836826 100 mg iv (Caucasian Patients) | BI 836826 100 mg iv (Korean Patients) | BI 836826 150 mg iv (Caucasian Patients) | BI 836826 200 mg iv (Caucasian Patients)
Number analyzed (Participants) | 1 | 4 | 3 | 4 | 6 | 7 | 6 | 4 | 6 | 7
days | 352.00 [352.00 to 352.00] | 87.00 [47.00 to 116.00] | 81.00 [17.00 to 199.00] | 22.00 [12.00 to 36.00] | 85.00 [18.00 to 262.00] | 25.00 [23.00 to 38.00] | 200.00 [62.00 to 218.00] | 51.50 [39.50 to 88.50] | 34.00 [22.00 to 44.00] | 36.00 [19.00 to 52.00]

ADVERSE EVENTS:
Time Frame: From the first drug (BI 836826) administration to 8 weeks after the last administration, ie up to 134 days
Arm/Group | BI 836826 1 mg iv (Caucasian Patients) | BI 836826 3 mg iv (Caucasian Patients) | BI 836826 9 mg iv (Caucasian Patients) | BI 836826 25 mg iv (Caucasian Patients) | BI 836826 50 mg iv (Caucasian Patients) | BI 836826 50mg iv (Korean Patients) | BI 836826 100 mg iv (Caucasian Patients) | BI 836826 100 mg iv (Korean Patients) | BI 836826 150 mg iv (Caucasian Patients) | BI 836826 200 mg iv (Caucasian Patients)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/4 | 1/3 | 1/4 | 2/6 | 1/7 | 1/6 | 1/4 | 2/6 | 1/7
Serious Adverse Events (participants affected / at risk) | 0/1 | 3/4 | 2/3 | 1/4 | 5/6 | 4/7 | 5/6 | 3/4 | 3/6 | 5/7
Other Adverse Events (participants affected / at risk) | 1/1 | 4/4 | 3/3 | 4/4 | 6/6 | 7/7 | 6/6 | 4/4 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 836826 1 mg iv (Caucasian Patients) (N=1) | BI 836826 3 mg iv (Caucasian Patients) (N=4) | BI 836826 9 mg iv (Caucasian Patients) (N=3) | BI 836826 25 mg iv (Caucasian Patients) (N=4) | BI 836826 50 mg iv (Caucasian Patients) (N=6) | BI 836826 50mg iv (Korean Patients) (N=7) | BI 836826 100 mg iv (Caucasian Patients) (N=6) | BI 836826 100 mg iv (Korean Patients) (N=4) | BI 836826 150 mg iv (Caucasian Patients) (N=6) | BI 836826 200 mg iv (Caucasian Patients) (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pulmonary mycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 836826 1 mg iv (Caucasian Patients) (N=1) | BI 836826 3 mg iv (Caucasian Patients) (N=4) | BI 836826 9 mg iv (Caucasian Patients) (N=3) | BI 836826 25 mg iv (Caucasian Patients) (N=4) | BI 836826 50 mg iv (Caucasian Patients) (N=6) | BI 836826 50mg iv (Korean Patients) (N=7) | BI 836826 100 mg iv (Caucasian Patients) (N=6) | BI 836826 100 mg iv (Korean Patients) (N=4) | BI 836826 150 mg iv (Caucasian Patients) (N=6) | BI 836826 200 mg iv (Caucasian Patients) (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 3 | 1 | 1 | 2 | 1 | 1 | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 1 | 3 | 0 | 5 | 0 | 4 | 4
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 3 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 2 | 2 | 4 | 5 | 4 | 3 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 1 | 3 | 4 | 3 | 1 | 1 | 4
Aortic valve calcification (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 0 | 3
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 3
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 2 | 2 | 1 | 3 | 2 | 1 | 5
Drug intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 3 | 2 | 0 | 1
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 3
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Oedema (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema mucosal (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 2 | 2
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 4
Swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angular cheilitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug administration error (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 1 | 1 | 3 | 2 | 1 | 6
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 2 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 2
CD4 lymphocytes decreased (Investigations) | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 2
Cytomegalovirus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 2
Fluid imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2 | 2 | 0 | 0 | 1 | 3 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Listless (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 2 | 1 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 2
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-04-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT01403948/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT01403948/SAP_001.pdf